CLINICAL TRIAL: NCT01298193
Title: A Prospective, Open Label, Non-comparative Trial to Determine the Incidence of Chemotherapy-Induced Nausea and Vomiting (CINV) Associated With the Docetaxel-Cyclophosphamide Regimen in Early Breast Cancer Patients
Brief Title: Incidence of Chemotherapy-Induced Nausea and Vomiting Associated With Docetaxel-Cyclophosphamide in Early Breast Cancer.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2009-02; 2010-022689-29 (EudraCT Number)
Record Dates: First submitted 2011-02-11; First posted 2011-02-17 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Early-stage breast cancer patients
MeSH Terms: conditions — Breast Neoplasms | interventions — Aprepitant; Serotonin 5-HT3 Receptor Antagonists; Phenothiazines; Butyrophenones; Haloperidol; Droperidol; Benzamides; Metoclopramide; alizapride; Benzodiazepines; Adrenal Cortex Hormones; Domperidone

STUDY DESIGN:
Intervention Model Description: Patients that experiment emesis within the first cycle in spite of the administration of antiemetics, may opt to participate in a subsequent efficacy phase
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aprepitant (Experimental): Observational phase (first cycle):
  Day 0 (Dexamethasone 8mg) Day 1 (5-HT3 antagonist, Ondansetron: 8 mg x2, Granisetron: 1mg x2,Tropisetron: 5 mg, Dexamethasone 24 mg) + Chemotherapy (Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 ).
  Days 2 and 3 (Dexamethasone 16 mg).
  If not complete response:
  Efficacy phase (second cycle):
  Day 0 (Dexamethasone 8mg) Day 1 (Aprepitant: 125 mg,5-HT3 antagonist, Ondansetron: 8 mg x2, Granisetron: 1mg x2, Tropisetron: 5 mg, Dexamethasone 12 mg)+ Chemotherapy: Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 .
  Days 2 and 3 (Aprepitant: 1 capsule of 80 mg daily, Dexamethasone 8 mg).
  Interventions: Drug: Aprepitant

INTERVENTIONS:
Drug: Aprepitant — Efficacy phase (second cycle)
  Other Names: Rescue therapy:Patients may be provided with a prescription.; - 5-HT3 antagonists; - Phenothiazines.; - Butyrophenones (e.g., haloperidol or droperidol); - Benzamides (e.g., metoclopramide or alizapride); - Benzodiazepines; - Corticosteroids; - Domperidone

SUMMARY:
This is a prospective, multicenter, open label, non-comparative trial in Spain.

The primary objective of this study is to determine the complete response, defined as no vomiting and no use of rescue treatment, in women with early-stage breast cancer treated with one cycle of Docetaxel-Cyclophosphamide and active therapy for the prevention of CINV (Chemotherapy-induced nausea and vomiting) day 1, 5-hydroxytryptamine 3 (5-HT3) antagonist plus 3 days of dexamethasone. A second step (efficacy phase) is designed to examine the efficacy and tolerability of aprepitant in the second cycle among patients who failed to the previous CINV prevention treatment.

The study will focus on early-stage chemonaive breast cancer patients receiving docetaxel-cyclophosphamide and a 5-HT3 antagonist plus dexamethasone for the CINV prevention. The CINV incidence in those patients will be evaluated on the first cycle. All refractory patients, will be asked to participate in the second phase, where aprepitant on days 1, 2 and 3 will be added to their antiemetic regimen.

Assuming a drop out of 5%, 212 patients will be included in the study. It is anticipated that around 48 patients will enter the efficacy phase.

The duration of the study, from first patient visit to last patient visit will be approximately 21 months.

DETAILED DESCRIPTION:
Sample size We want to obtain an estimation of the percent of the patients that we assume won't have a response to the treatment against vomiting. Reviewing bibliography, we think that the percent is approximately 25%.

We are going to obtain an estimation of this percent with an accuracy of +/- 6%, with a bilateral confidence level of 95% bilateral. Whit all this premises it would be needed 201 patients.

Assuming a drop out of 5%, 212 patients will be included in the study.

A maximum of 212 patients will be included in the trial. It is anticipated that around 48 patients will enter the efficacy phase.

APPROXIMATE DURATION OF THE STUDY. Inclusion period: 18 months approximately. Estimated follow-up: December 2012 Estimated date of end of study: June 2013

ELIGIBILITY:
Inclusion Criteria:

1. Female patient ≥ 18 years of age.
2. Patient has a histological confirmed early-stage (I to III) breast cancer.
3. Patient is able to understand study procedures and agrees to participate in the study by giving written informed consent.
4. Patient is naive to moderate or highly emetogenic chemotherapy per "Hesketh" criteria.
5. Patient is scheduled to receive of chemotherapy with Docetaxel-Cyclophosphamide (Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2) administered every 21 days.
6. Patient has a predicted life expectancy ≥ 4 months.
7. Functional State 0-1 Eastern Cooperative Oncology Group (ECOG) Scale (see Appendix 12.2).
8. Patient has an adequate organ function including the following:

   * Bone marrow reserve: Absolute Neutrophil Count >1500/mm3 and white blood cell (WBC) count >3000/mm3; Platelet Count >100.000/mm3
   * Hepatic: aspartate aminotransferase (AST) <2.5 x upper limit of normal; alanine aminotransferase (ALT) <2.5 x upper limit of normal; Bilirubin within the normal limit.
   * Renal: Creatinine <1.5 x upper limit of normal.
9. Premenopausal female patients must demonstrate a negative serum and/or urine pregnancy test within 3 days of study drug administration, and agree to use a double-barrier form of contraception for at least 14 days prior to, throughout and for at least 14 days following the last dose of study medication. Women taking oral contraceptive agents must agree to add a barrier form of contraception. Abstinence is also considered an acceptable form of contraception. (Note: A female patient who is not of reproductive potential is eligible without requiring the use of contraception. A female patient who is not of reproductive potential is defined as one who has either: 1) reached natural menopause (defined as 6 months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels in the postmenopausal range as determined by the laboratory, or 12 months of spontaneous amenorrhea); 2) 6 weeks post surgical bilateral oophorectomy with or without hysterectomy; or 3) bilateral tubal ligation.)
10. Patient is able to read, understand and complete study questionnaires.

Exclusion Criteria:

1. Patient is scheduled to receive any chemotherapy treatment different to the Docetaxel-Cyclophosphamide chemotherapy.
2. Patient has received or will receive radiation therapy to the abdomen, chest or pelvis in the month prior to the study enter.
3. Patient has vomited in the 24 hours prior to Treatment Day 1.
4. Patient has a history of treatment with emetogenic chemotherapy of moderate or high level per "Hesketh" (classification of emetogenic chemotherapy agents).
5. Patient has an active infection (e.g., pneumonia) or any uncontrolled disease (e.g., diabetic ketoacidosis, gastrointestinal obstruction) except for malignancy which, in the opinion of the investigator, might confound the results of the study or pose unwarranted risk.
6. Patient currently uses any illicit drugs, including marijuana, or has current evidence of alcohol abuse as determined by the investigator.
7. Patient is mentally incapacitated or has a significant emotional or psychiatric disorder that, in the opinion of the investigator, precludes study entry.
8. Patient has a history of any illness that, in the opinion of the investigator, might confound the results of the study or pose unwarranted risk.
9. Patient has a history of hypersensitivity to aprepitant, 5-HT3 antagonists, or dexamethasone.
10. Patient is pregnant or breast feeding.
11. Patient has participated in a study with aprepitant or has taken a non approved (investigational) drug within the last 4 weeks.
12. Patient is taking systemic corticosteroid therapy at any dose; topical and inhaled corticosteroids are permitted.
13. Patient is taking, or will be taking within 28 days of Day 1 of cycle 2 (cycle in which patients will start taking aprepitant) the following CYP3A4 inducers:

    * phenytoin or carbamazepine
    * barbiturates
    * rifampicin or rifabutin
    * St. John's Wort
14. Patient is taking, or will be taking within 7 days of Day 1 of cycle 2 the following CYP3A4 substrates:

    * terfenadine
    * cisapride
    * astemizole
    * pimozide
15. Patient is taking, or will be taking within the 7 days of Day 1 of cycle 2 the following CYP3A4 inhibitors:

    * clarithromycin
    * ketoconazole, itraconazole
16. Patient will be taking an antiemetic within 48 hours of Day 1 of cycle 2. Prohibited antiemetics include:

    * 5-HT3 antagonists (ondansetron, granisetron, dolasetron, tropisetron or palonosetron)
    * phenothiazines (e.g., prochlorperazine, fluphenazine, perphenazine, thiethylperazine, or chlorpromazine)
    * butyrophenones (e.g., haloperidol or droperidol)
    * benzamides (e.g., metoclopramide or alizapride)
    * domperidone
    * cannabinoids
    * herbal therapies with potential antiemetic properties
    * scopolamine
    * cyclizine
17. Patient has used benzodiazepines or opiates, except for single daily doses of triazolam, temazepam or midazolam in the 48 hours prior to Day 1 of cycle 2. Continuation of chronic benzodiazepines or opiate therapy is permitted provided it was initiated at least 48 hours before enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Universitario Arnau de Vilanova; Study Director, Study Director — Fundación Hospital Alcorcón
Locations (13):
- Spain (13):
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Oncológico de Galicia, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Complejo Hospitalario Xeral-Calde, Lugo
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Result] Llombart-Cussac A, Ramos M, Dalmau E, Garcia-Saenz JA, Gonzalez-Farre X, Murillo L, Calvo L, Morales S, Caranana V, Gonzalez A, Fernandez-Morales LA, Moreno F, Casas MI, Angulo Mdel M, Camara MC, Garcia-Mace AI, Carrasco E, Jara-Sanchez C. Incidence of chemotherapy-induced nausea and vomiting associated with docetaxel and cyclophosphamide in early breast cancer patients and aprepitant efficacy as salvage therapy. Results from the Spanish Breast Cancer Group/2009-02 study. Eur J Cancer. 2016 May;58:122-9. doi: 10.1016/j.ejca.2016.01.015. Epub 2016 Mar 17. PMID 26994459
- See also: Sponsor's website — http://www.geicam.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The investigator registered all the selected patients before the start of the treatment.
  Once it was verified that the selection criteria were complied with, the investigator sent the previously completed randomization sheet by fax to Spanish Breast Cancer Research Group (GEICAM).
  Recruitment period: From May-2011 to 31-Jan-13.
Groups:
- Aprepitant: Observational phase (first cycle):
  Day 0: Dexamethasone 8mg Day 1: 5-HydroxyTryptamine 3 (5-HT3) antagonist, Ondansetron: 8 mg x2, Granisetron: 1mg x2,Tropisetron: 5 mg, Dexamethasone 24 mg.
  • Chemotherapy: Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 Days 2 and 3: Dexamethasone 16 mg.
  Patients that experiment emesis within the first cycle in spite of the administration of antiemetics goes to efficacy phase (Second cycle):
  Day 0: dexamethasone oral (8 mg Day 1: iv/oral* 5-hydroxytryptamine 3 [5-HT3] + dexamethasone oral (4mg x 3) + aprepitant oral 125mg
  • Chemotherapy: Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 Day 2 and 3: dexamethasone oral (4mg x 2) + oral aprepitant 80mg
Period: Observational Phase (First Cycle)
Arm/Group | Aprepitant
Started | 212
Completed | 185 (From these 185 completed patients, only 24 experiment emesis on Cycle 1 (NCR) (efficacy phase).)
Not Completed | 27
Not completed — Withdrawal by Subject | 2
Not completed — Received TC at a different dose | 16
Not completed — previous emetogenic chemotherapy | 9
Period: Efficacy Phase (Second Cycle)
Arm/Group | Aprepitant
Started | 24
Completed | 23
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: From May 2011 to March 2013, 212 Early Breast Cancer (EBC) patients from 12 sites in Spain were recruited.
Groups:
- Aprepitant: Observational phase (first cycle):
  Day 0 (Dexamethasone 8mg) Day 1 (5-HT3 antagonist, Ondansetron: 8 mg x2, Granisetron: 1mg x2,Tropisetron: 5 mg, Dexamethasone 24 mg).
  • Chemotherapy: Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 Days 2 and 3 (Dexamethasone 16 mg).
  Efficacy phase (second cycle):
  Day 0 (Dexamethasone 8mg) Day 1 (Aprepitant: 125 mg,5-HT3 antagonist, Ondansetron: 8 mg x2, Granisetron: 1mg x2, Tropisetron: 5 mg, Dexamethasone 12 mg).
  Chemotherapy: Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 Days 2 and 3 (Aprepitant: 1 capsule of 80 mg daily, Dexamethasone 8 mg).
  Aprepitant: Efficacy phase (second cycle)
Arm/Group | Aprepitant
Number analyzed (Participants) | 212
Age, Continuous [Median (Full Range); unit: years] | 57 [34 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 201
  Hispanic | 9
  Asian | 1
  Arab | 1
Eastern Cooperative Oncology Group (ECOG) status [Count of Participants; unit: Participants] — ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death. 0 - Asymptomatic
  1. - Symptomatic but completely ambulatory
  2. - Symptomatic, <50% in bed during the day
  3. - Symptomatic, >50% in bed, but not bedbound
  4. - Bedbound
  5. - Death
  Participants
    ECOG 0 | 185
    ECOG 1 | 19
    Missing | 8
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 62
  Postmenopausal | 150
Drink alcohol [Count of Participants; unit: Participants]
  Yes | 37
  No | 168
  Not available | 7
Regularly dizziness [Count of Participants; unit: Participants]
  Yes | 22
  No | 176
  Not available | 14
Morning nausea during pregnancy [Count of Participants; unit: Participants]
  Yes | 45
  No | 142
  Not available | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR)
Description: Complete response is defined as no vomiting and no use of rescue treatment within the first cycle of Docetaxel-Cyclophosphamide for the treatment of early-stage breast cancer patients. A vomiting episode is defined as one or more episodes of emesis (expulsion of stomach contents through the mouth) or retches (an attempt to vomit that is not productive of stomach contents). Distinct vomiting episodes are, by definition, separated by the absence of emesis and retching for at least 1 minute. The timing (date and time) of each vomiting episode will be recorded by the patient in each cycle diary at the time of occurrence. Assessments of efficacy will begin at the initiation of chemotherapy infusion (0 hours) until the morning of Day 6 (approximately 120 hours) after chemotherapy during 1-2 cycles.
Time Frame: Up to 21 days after cycle 1 of chemotherapy treatment
Population: 27 patients were excluded from the main analysis: 16 received docetaxel and cyclophosphamide (TC) at a different dose from that in the protocol, 9 had received previous emetogenic chemotherapy and 2 withdrew study consent before receiving TC.
Measure: Count of Participants; unit: Participants
Groups:
- Observational Phase (First Cycle):: Observational phase (first cycle):
  Day 0 (Dexamethasone 8mg) Day 1 (5-hydroxytryptamine 3 [5-HT3] antagonist, Ondansetron: 8 mg x2, Granisetron: 1mg x2,Tropisetron: 5 mg, Dexamethasone 24 mg).
  • Chemotherapy: Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 Days 2 and 3 (Dexamethasone 16 mg).
Arm/Group | Observational Phase (First Cycle):
Number analyzed (Participants) | 185
Participants | 161

2. Secondary Outcome: Number of Participants With Complete Response (CR) in Cycle 2 for Patient Without Complete Response in Cycle 1
Description: To evaluate in cycle 2 the efficacy of aprepitant (days 1, 2 and 3) as secondary prevention in patients without complete response in cycle 1. A vomiting episode is defined as one or more episodes of emesis (expulsion of stomach contents through the mouth) or retches (an attempt to vomit that is not productive of stomach contents). Distinct vomiting episodes are, by definition, separated by the absence of emesis and retching for at least 1 minute. The timing (date and time) of each vomiting episode will be recorded by the patient in each cycle diary at the time of occurrence. Assessments of efficacy will begin at the initiation of chemotherapy infusion (0 hours) until the morning of Day 6 (approximately 120 hours) after chemotherapy during 1-2 cycles.
Time Frame: Up to cycle 2, and average of 6 weeks
Population: Of the 185 evaluable patients, 161 achieved CR, so who participated in this outcome were 24 patients who experienced non-complete response (NCR).
Measure: Count of Participants; unit: Participants
Groups:
- Aprepitant NCR: Patients that experiment emesis within the first cycle in spite of the administration of antiemetics goes to efficacy phase (Second cycle):
  Day 0: dexamethasone oral (8 mg Day 1: iv/oral* 5-hydroxytryptamine 3 [5-HT3] + dexamethasone oral (4mg x 3) + aprepitant oral 125mg
  • Chemotherapy: Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 Day 2 and 3: dexamethasone oral (4mg x 2) + oral aprepitant 80mg
Arm/Group | Aprepitant NCR
Number analyzed (Participants) | 24
Participants | 12

3. Secondary Outcome: Number of Participants With Treatment Related Adverse Events (AE) at Cycle 2
Description: Events are related to the primary end point, they were collected only in the diary during the period of diary data collection (Day 1 to the morning of Day 6) for the cycle 2, unless they meet the definition of a serious adverse event.
Time Frame: Cycle 2, and average of 3 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Aprepitant NCR
Number analyzed (Participants) | 24
Participants | 0

4. Secondary Outcome: Total Impact of Chemotherapy-Induced Nausea and Vomiting on Daily Life by the Functional Living Index-Emesis Questionnaire in Cycle 1
Description: To determine the incidence of Chemotherapy-Induced Nausea and Vomiting associated with the Docetaxel-Cyclophosphamide regimen in early breast cancer patients, a Functional Living Index-Emesis (FLIE) questionnaire was collected on treatment Day 1 (prior to initiation of chemotherapy) and Day 6, which referenced the entire treatment period since the initiation of chemotherapy for non clinical responders (NCR) against clinical responders (CR).
  The FLIE questionnaire is a validated, patient-reported instrument to measure the impact of Chemotherapy-Induced Nausea and Vomiting on daily life. There are 18 items, each on a 7-point scale. Results are reported as a total score. For the purposes of this study, higher scores indicate less impairment on daily life as a result of nausea or vomiting (better outcome) (Maximum 126, Minimum 18).
Time Frame: Up to day 6
Population: From 212 patients randomized, 27 were not evaluable patients. From the rest 185, 161 presented CR, and 24 a NCR.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Aprepitant: Observational phase (first cycle):
  Day 0 (Dexamethasone 8mg) Day 1 (5-hydroxytryptamine 3 [5-HT3] antagonist, Ondansetron: 8 mg x2, Granisetron: 1mg x2,Tropisetron: 5 mg, Dexamethasone 24 mg).
  • Chemotherapy: Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 Days 2 and 3 (Dexamethasone 16 mg).
  Patients that experiment emesis within the first cycle in spite of the administration of antiemetics goes to efficacy phase (Second cycle):
  Day 0: dexamethasone oral (8 mg Day 1: iv/oral* 5-hydroxytryptamine 3 [5-HT3] + dexamethasone oral (4mg x 3) + aprepitant oral 125mg
  • Chemotherapy: Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 Day 2 and 3: dexamethasone oral (4mg x 2) + oral aprepitant 80mg
Arm/Group | Aprepitant
Number analyzed (Participants) | 185
score on a scale
  Cycle 1 pre-chemotherapy NCR patients: number analyzed (Participants) | 24
  Cycle 1 pre-chemotherapy NCR patients | 43.7 [36.36 to 51.05]
  Cycle 1 post-chemotherapy NCR patients: number analyzed (Participants) | 24
  Cycle 1 post-chemotherapy NCR patients | 59.2 [50.59 to 67.75]
  Cycle 1 pre-chemotherapy CR patients: number analyzed (Participants) | 161
  Cycle 1 pre-chemotherapy CR patients | 42.5 [39.99 to 44.94]
  Cycle 1 post-chemotherapy CR patients: number analyzed (Participants) | 161
  Cycle 1 post-chemotherapy CR patients | 44.22 [42.04 to 46.79]

5. Secondary Outcome: Impact of Chemotherapy-Induced Nausea on Daily Life by the Functional Living Index-Emesis Questionnaire in Cycle 1
Description: To determine the incidence of nausea associated with the Docetaxel-Cyclophosphamide regimen in early breast cancer patients, a Functional Living Index-Emesis (FLIE) questionnaire was collected on treatment Day 1 (prior to initiation of chemotherapy) and Day 6, which referenced the entire treatment period since the initiation of chemotherapy for non clinical responders (NCR) against clinical responders (CR).
  The FLIE questionnaire is a validated, patient-reported instrument to measure the impact of Chemotherapy-Induced Nausea and vomiting on daily life. There are 9 nausea-related items, each on a 7-point scale. Results are reported as a nausea score. For the purposes of this study, higher scores indicate less impairment on daily life as a result of nausea (better outcome) (Maximum 63, Minimum 9).
Time Frame: Up to day 6
Population: From 212 patients randomized, 27 were not evaluable patients. From the rest 185, 161 presented CR, and 24 a NCR.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aprepitant
Number analyzed (Participants) | 185
score on a scale
  Cycle 1 pre-chemotherapy NCR patients: number analyzed (Participants) | 24
  Cycle 1 pre-chemotherapy NCR patients | 19.85 [16.23 to 23.46]
  Cycle 1 post-chemotherapy NCR patients: number analyzed (Participants) | 24
  Cycle 1 post-chemotherapy NCR patients | 31.73 [26.56 to 36.89]
  Cycle 1 pre-chemotherapy CR patients: number analyzed (Participants) | 161
  Cycle 1 pre-chemotherapy CR patients | 18.93 [17.76 to 20.10]
  Cycle 1 post-chemotherapy CR patients: number analyzed (Participants) | 161
  Cycle 1 post-chemotherapy CR patients | 20.27 [19.12 to 21.42]

6. Secondary Outcome: Impact of Chemotherapy-Induced Vomiting on Daily Life by the Functional Living Index-Emesis Questionnaire in Cycle 1
Description: To determine the incidence of vomiting associated with the Docetaxel-Cyclophosphamide regimen in early breast cancer patients, a Functional Living Index-Emesis (FLIE) questionnaire was collected on treatment Day 1 (prior to initiation of chemotherapy) and Day 6, which referenced the entire treatment period since the initiation of chemotherapy for non clinical responders (NCR) against clinical responders (CR).
  The FLIE questionnaire is a validated, patient-reported instrument to measure the impact of vomiting on daily life. There are 9 vomiting-related items, each on a 7-point scale. Results are reported as a vomiting score. For the purposes of this study, higher scores indicate less impairment on daily life as a result of vomiting (better outcome) (Maximum 63, Minimum 9).
Time Frame: Up to day 6
Population: From 212 patients randomized, 27 were not evaluable patients. From the rest 185, 161 presented CR, and 24 a NCR.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aprepitant
Number analyzed (Participants) | 185
score on a scale
  Cycle 1 pre-chemotherapy NCR patients: number analyzed (Participants) | 24
  Cycle 1 pre-chemotherapy NCR patients | 23.86 [19.84 to 27.89]
  Cycle 1 post-chemotherapy NCR patients: number analyzed (Participants) | 24
  Cycle 1 post-chemotherapy NCR patients | 27.46 [22.01 to 32.88]
  Cycle 1 pre-chemotherapy CR patients: number analyzed (Participants) | 161
  Cycle 1 pre-chemotherapy CR patients | 23.53 [22.07 to 25]
  Cycle 1 post-chemotherapy CR patients: number analyzed (Participants) | 161
  Cycle 1 post-chemotherapy CR patients | 24.15 [22.76 to 25.54]

7. Secondary Outcome: Total Impact of Chemotherapy-Induced Nausea and Vomiting on Daily Life by the Functional Living Index-Emesis Questionnaire in Cycle 2
Description: To determine the total incidence of Chemotherapy-Induced Nausea and Vomiting associated with the Docetaxel-Cyclophosphamide regimen in early breast cancer patients, a Functional Living Index-Emesis (FLIE) questionnaire was collected on treatment Day 1 (prior to initiation of chemotherapy) and Day 6, which referenced the entire treatment period since the initiation of chemotherapy for non clinical responders (NCR) against clinical responders (CR).
  The FLIE questionnaire is a validated, patient-reported instrument to measure the impact of Chemotherapy-Induced Nausea and Vomiting on daily life. There are 18 items, each on a 7-point scale. Results are reported as a total score. For the purposes of this study, higher scores indicate less impairment on daily life as a result of nausea or vomiting (better outcome) (Maximum 126, Minimum 18).
Time Frame: Up to day 6
Population: During cycle 2, only 23 patients completed the FLIE questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aprepitant NCR
Number analyzed (Participants) | 23
score on a scale
  Cycle 2 pre-chemotherapy NCR patients: number analyzed (Participants) | 11
  Cycle 2 pre-chemotherapy NCR patients | 37.8 [25.74 to 49.86]
  Cycle 2 post-chemotherapy NCR patients: number analyzed (Participants) | 11
  Cycle 2 post-chemotherapy NCR patients | 64.4 [52.07 to 76.64]
  Cycle 2 pre-chemotherapy CR patients: number analyzed (Participants) | 12
  Cycle 2 pre-chemotherapy CR patients | 43.28 [30.20 to 56.36]
  Cycle 2 post-chemotherapy CR patients: number analyzed (Participants) | 12
  Cycle 2 post-chemotherapy CR patients | 47.7 [43.7 to 51.75]

8. Secondary Outcome: Impact of Chemotherapy-Induced Nausea on Daily Life by the Functional Living Index-Emesis Questionnaire in Cycle 2
Description: To determine the incidence of Nausea associated with the Docetaxel-Cyclophosphamide regimen in early breast cancer patients, a Functional Living Index-Emesis (FLIE) questionnaire was collected on treatment Day 1 (prior to initiation of chemotherapy) and Day 6, which referenced the entire treatment period since the initiation of chemotherapy for non clinical responders (NCR) against clinical responders (CR).
  The FLIE questionnaire is a validated, patient-reported instrument to measure the impact of Nausea on daily life. There are 9 items, each on a 7-point scale. Results are reported as a nausea score. For the purposes of this study, higher scores indicate less impairment on daily life as a result of nausea (better outcome) (Maximum 63, Minimum 9).
Time Frame: Up to day 6
Population: During cycle 2, only 23 patients completed the FLIE questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aprepitant NCR
Number analyzed (Participants) | 23
score on a scale
  Cycle 2 pre-chemotherapy NCR patients: number analyzed (Participants) | 11
  Cycle 2 pre-chemotherapy NCR patients | 17.71 [11.07 to 24.35]
  Cycle 2 post-chemotherapy NCR patients: number analyzed (Participants) | 11
  Cycle 2 post-chemotherapy NCR patients | 36.16 [28.26 to 44.07]
  Cycle 2 pre-chemotherapy CR patients: number analyzed (Participants) | 12
  Cycle 2 pre-chemotherapy CR patients | 19.57 [13.66 to 25.48]
  Cycle 2 post-chemotherapy CR patients: number analyzed (Participants) | 12
  Cycle 2 post-chemotherapy CR patients | 24.30 [20.35 to 28.25]

9. Secondary Outcome: Impact of Chemotherapy-Induced Vomiting on Daily Life by the Functional Living Index-Emesis Questionnaire in Cycle 2
Description: To determine the incidence of vomiting associated with the Docetaxel-Cyclophosphamide regimen in early breast cancer patients, a Functional Living Index-Emesis (FLIE) questionnaire was collected on treatment Day 1 (prior to initiation of chemotherapy) and Day 6, which referenced the entire treatment period since the initiation of chemotherapy for non clinical responders (NCR) against clinical responders (CR).
  The FLIE questionnaire is a validated, patient-reported instrument to measure the impact of vomiting on daily life. There are 9 items, each on a 7-point scale. Results are reported as a vomiting score. For the purposes of this study, higher scores indicate less impairment on daily life as a result of vomiting (better outcome) (Maximum 63, Minimum 9).
Time Frame: Up to day 6
Population: During cycle 2, only 23 patients completed the FLIE questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aprepitant NCR
Number analyzed (Participants) | 23
score on a scale
  Cycle 2 pre-chemotherapy NCR patients: number analyzed (Participants) | 11
  Cycle 2 pre-chemotherapy NCR patients | 20.09 [12.82 to 27.36]
  Cycle 2 post-chemotherapy NCR patients: number analyzed (Participants) | 11
  Cycle 2 post-chemotherapy NCR patients | 28.19 [21.91 to 34.47]
  Cycle 2 pre-chemotherapy CR patients: number analyzed (Participants) | 12
  Cycle 2 pre-chemotherapy CR patients | 23.71 [16.40 to 31.02]
  Cycle 2 post-chemotherapy CR patients: number analyzed (Participants) | 12
  Cycle 2 post-chemotherapy CR patients | 23.43 [17.55 to 29.30]

ADVERSE EVENTS:
Time Frame: Through study treatment, average of 6 weeks
Description: This section includes related and no related Adverse Events and Serious Adverse Events. There are not adverse events related to aprepitant treatment in cycle 2.
Groups:
- Observational Phase (First Cycle):: Day 0 (Dexamethasone 8mg) Day 1 (5-HT3 antagonist, Ondansetron: 8 mg x2, Granisetron: 1mg x2,Tropisetron: 5 mg, Dexamethasone 24 mg).
  • Chemotherapy: Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 Days 2 and 3 (Dexamethasone 16 mg).
- Efficacy Phase (Second Cycle):: Day 0 (Dexamethasone 8mg) Day 1 (Aprepitant: 125 mg,5-HT3 antagonist, Ondansetron: 8 mg x2, Granisetron: 1mg x2, Tropisetron: 5 mg, Dexamethasone 12 mg).
  Chemotherapy: Docetaxel 75mg/m2 and Cyclophosphamide 600mg/m2 Days 2 and 3 (Aprepitant: 1 capsule of 80 mg daily, Dexamethasone 8 mg).
Arm/Group | Observational Phase (First Cycle): | Efficacy Phase (Second Cycle):
All-Cause Mortality (participants affected / at risk) | 1/185 | 0/24
Serious Adverse Events (participants affected / at risk) | 31/185 | 0/24
Other Adverse Events (participants affected / at risk) | 47/185 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Phase (First Cycle): (N=185) | Efficacy Phase (Second Cycle): (N=24)
Anemic Shock (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 13 (13) | 0 (0) — Grade 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Colon Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) — Grade 4
Lower Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3
Erythema with pruritus and skin lessions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Grade 4
Enterocollitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Grade 3
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Grade 4
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Grade 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Phase (First Cycle): (N=185) | Efficacy Phase (Second Cycle): (N=24)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) — Grade 3
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) — Grade 3
Nausea (Gastrointestinal disorders) | 14 (14) | 4 (4) — Grade 2
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) — Grade 2
Nausea (Gastrointestinal disorders) | 14 (14) | 12 (12) — Grade 1
Vomiting (Gastrointestinal disorders) | 13 (13) | 3 (3) — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No